CLINICAL TRIAL: NCT00165841
Title: A Double-Blind, Placebo-Controlled Study of Rabeprazole 20 mg Maintenance Intermittent Therapy Following Acute Treatment in Patients Wth Symptomatic Gastroesophageal Reflux Disease
Brief Title: Maintenance Intermittent Therapy for Symptomatic GERD Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Yufang Lu, Study Director, Eisai Medical Research Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E3810-A001-203
Record Dates: First submitted 2005-09-13; First posted 2005-09-14 (Estimated); Results first posted 2009-12-03 (Estimated); Last update posted 2013-05-20 (Estimated); Status verified 2009-12

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: non-erosive symptomatic GERD; GERD
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Rabeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Rabeprazole 20 mg
- Rabeprazole 20 mg (Experimental)
  Interventions: Drug: Rabeprazole 20 mg

INTERVENTIONS:
Drug: Rabeprazole 20 mg — rabeprazole sodium tablet 20 mg once daily
  Other Names: rabeprazole

SUMMARY:
The purpose of this study to determine the efficacy of 20 mg of rabeprazole given as a maintenance intermittent therapy following acute treatment for Symptomatic Gastroesophageal Reflux Disease (s-GERD).

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female patients, 18 to 65 years of age.
2. If female, not of childbearing potential by reason of surgery, radiation or menopause, or of childbearing potential, but using an approved method of contraception since the last menstrual period, for example, intrauterine device (IUD), implant, double barrier method, or oral contraceptives for at least one cycle. Females of childbearing potential must have a negative urine pregnancy test before medication is dispensed.
3. Patients must report a minimum three-month history of GERD symptoms. GERD symptoms are defined as heartburn with or without regurgitation or other associated GERD symptoms.
4. Patients must have at least 4 days with heartburn per week in each of the 2 weeks prior to Screening.
5. Patients must have no esophagitis, with no proton pump inhibitors (PPIs, prescription or OTC), H2 blockers (prescription or OTC) or prokinetics within 14 days, prior to the endoscopy.

Key Exclusion Criteria:

1. Evidence of significant hepatic, renal, respiratory, endocrine, hematologic, neurologic, psychiatric or cardiovascular system abnormalities, unless the Sponsor and Investigator agree that the nature and severity of any abnormality is unlikely to interfere with the conduct of the study, the interpretation of study results, or the health of the patient during the study.
2. Females must not be pregnant, lactating or have a positive urine eta human chorionic gonadotropin (B-hCG) laboratory result.
3. Patients with a history of allergy or sensitivity to proton pump inhibitors or to their inactive ingredients.
4. Patients with known gastric ulcer, duodenal ulcer, infectious or inflammatory conditions of the small or large intestine, malabsorption syndromes, obstruction, a history of gastrointestinal malignancy, or prior gastric or intestinal surgery (including vagotomy).
5. Patients who have a history of Barrett's esophagus, esophageal stricture, or pyloric stenosis.
6. Patients with a history of endoscopically-proven esophagitis any time in the past.
7. Patients who have taken proton pump inhibitors (PPIs, prescription or OTC), H2 blockers (prescription or OTC) or prokinetics within 14 days, prior to Screening endoscopy, or any of these medications within 7 days prior to the single-blind placebo run-in period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2004-10; Primary Completion 2005-12 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yufang Lu, Study Director — Eisai Inc.
Locations (1):
- Quality Care Medical Center Inc., Vista, California, United States

REFERENCES:
- [Derived] Fass R, Delemos B, Nazareno L, Kao R, Xiang J, Lu Y. Clinical trial: maintenance intermittent therapy with rabeprazole 20 mg in patients with symptomatic gastro-oesophageal reflux disease - a double-blind, placebo-controlled, randomized study. Aliment Pharmacol Ther. 2010 May;31(9):950-60. doi: 10.1111/j.1365-2036.2010.04254.x. Epub 2010 Feb 2. PMID 20132154

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was recruited at 47 centers in the US during the period of 7-Oct-2004 and 12-Dec-2005.
Pre-assignment Details: After enrollment and before randomization (treatment assignment), there was a 2-week placebo run-in phase followed by a 4-week open-label Acute Phase during which subjects were treated with rabeprazole 20 mg once daily for the treatment of heartburn. Note the below participant flow is based on Safety Population (total 200 subjects).
Groups:
- Rabeprazole 20 mg; Placebo: Orally, once daily for 7- to 14-day courses intermittently during the 6-month Double-blind Maintenance Treatment Phase.
Period: Overall Study
Arm/Group | Rabeprazole 20 mg | Placebo
Started | 103 | 97
Completed | 73 | 35
Not Completed | 30 | 62
Not completed — Adverse Event | 2 | 3
Not completed — Lack of Efficacy | 6 | 33
Not completed — Lost to Follow-up | 4 | 4
Not completed — Withdrawal by Subject | 7 | 8
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Violation | 6 | 8
Not completed — Other | 3 | 5
Not completed — Medication Noncompliance | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Rabeprazole 20 mg; Placebo: Orally, once daily for 7 to 14-day courses intermittently during the 6-month Maintenance Treatment Phase (ITT population).
- Total: Total of all reporting groups
Arm/Group | Rabeprazole 20 mg | Placebo | Total
Number analyzed (Participants) | 96 | 91 | 187
Age Continuous [Mean (Standard Deviation); unit: years] | 46.0 (11.67) | 46.6 (11.69) | 46.3 (11.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 59 | 123
  Male | 32 | 32 | 64
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 10 | 19
  White | 74 | 64 | 138
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 12 | 16 | 28

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Heartburn-free Days (24-hour Periods) During the 6-month Maintenance Treatment Phase (ITT Population).
Description: The percentage of heartburn-free days during the 6-month Maintenance Treatment Phase in patients treated with rabeprazole 20 mg compared to patients who received placebo in the ITT Population. Heartburn-free day was defined as no heartburn in both the daytime and nighttime period on a given day. Note a total 388 subjects were enrolled at the beginning of Acute Phase and 200 subjects were enrolled into the double-blind 6-month maintenance treatment phase.
Time Frame: 6 months double-blind maintenance phase
Population: Intent-to-treat (ITT) population, total 187 subjects, was used for efficacy analyses. Safety population (total 200 subjects) was used for safety analysis and participant flow.
Measure: Mean (Standard Deviation); unit: Percentage of Days
Arm/Group | Rabeprazole 20 mg | Placebo
Number analyzed (Participants) | 96 | 91
Percentage of Days | 82.58 (14.39) | 62.17 (29.93)
Statistical Analysis 1: Comparison: Rabeprazole 20 mg vs Placebo; Efficacy analyses were based on the intent-to-treat (ITT) population, which was comprised of all patients in the safety-evaluable population who had a baseline and ≥1 post-randomization primary efficacy endpoint evaluation and who had received ≥1 dose of study medication during the maintenance phase; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — p-value was adjusted for multiple comparisons; The primary analysis was on the ITT population using all observed data collected from Day 1 of the maintenance phase until the endpoint

2. Secondary Outcome: The Percent of Heartburn-free Daytime Period During the 6-month Maintenance Treatment Phase
Description: The percentage of heartburn-free daytime period is presented cumulatively including all data collected during the 6-month Maintenance Phase
Time Frame: 6-month maintenance phase
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: %

3. Secondary Outcome: The Percent of Heartburn-free Nighttime Period During the 6-month Maintenance Treatment Phase
Description: The percentage of heartburn-free nighttime period is presented cumulatively including all data collected during the 6-month
Time Frame: 6-month maintenance phase
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: %

ADVERSE EVENTS:
Time Frame: 6 month maintenance phase
Description: Safety population (total 200 subjects) was used for safety analysis and participant flow.
Arm/Group | Rabeprazole 20 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 2 | 2
Other Adverse Events (participants affected / at risk) | 38 | 36
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Rabeprazole 20 mg | Placebo
Gallstone pancreatitis (Gastrointestinal disorders) | 0/103 (0) | 1/97 (1)
Pneumonia (Infections and infestations) | 0/103 (0) | 1/97 (1)
Chest pain (General disorders) | 1/103 (1) | 0/97 (0)
Schizoaffective disorder/depression (Nervous system disorders) | 1/103 (1) | 0/97 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Rabeprazole 20 mg | Placebo
Diarrhea (Gastrointestinal disorders) | 7/103 | 1/97
Erosive gastritis (Gastrointestinal disorders) | 2/103 | 4/97
Hiatus hernia (Gastrointestinal disorders) | 6/103 | 4/97
Nausea (Gastrointestinal disorders) | 5/103 | 3/97
Esophageal erosion (Gastrointestinal disorders) | 2/103 | 6/97
Esophagitis (Gastrointestinal disorders) | 4/103 | 5/97
Viral gastroenteritis (Infections and infestations) | 0/103 | 4/97
Sinusitis (Infections and infestations) | 2/103 | 4/97
Headache (Nervous system disorders) | 5/103 | 3/97
Cough (Respiratory, thoracic and mediastinal disorders) | 5/103 | 2/97

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other